CLINICAL TRIAL: NCT02821611
Title: Physical Therapist Doctoral Student Stress Levels and Management Through Meditation
Brief Title: Student Stress Levels and Management Through Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Northridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1314-136-b
Record Dates: First submitted 2016-04-18; First posted 2016-07-01 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Stress, Psychological
Keywords: Student Stress; Meditation; Sleep Quality; Blood Pressure
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation Group (Experimental): Participants in the experimental group are practicing a mantra-based meditation twice daily for 20 minutes over the 8 week intervention period to reduce stress and blood pressure and enhance quality of sleep.
  Interventions: Behavioral: Meditation Group
- Control Group (No Intervention): Control group participants will continue their normal activities and not add any form of meditation during the study period.

INTERVENTIONS:
Behavioral: Meditation Group — twice daily 20 minute mantra-based meditation practice for 8 weeks
  Arms: Meditation Group

SUMMARY:
The professional program in Physical Therapy is rigorous and demanding on students, resulting in high levels of fatigue, stress, and sleep disturbance that can impact student performance and wellbeing. This project seeks to investigate ways to reduce student stress, monitor their quality of sleep and possibly enhance their learning through the practice of meditation.

DETAILED DESCRIPTION:
Utilizing a randomized controlled study design, a cohort of doctoral students in their first year of physical therapist education will undergo an 8 week intervention of a mantra-based Meditation (twice daily 20 minutes) with pre and post measures of blood pressure, sleep hygiene via the Pittsburgh Sleep Quality Index (PSQI) and stress surveys, including Perceived Stress Scale (PSS) and Visual Analogue Scale for stress (VAS), as well as daily logs of sleep to assess sleep quality.

As many as 32 students (total number in cohort) per year may participate with 1/2 serving as controls and 1/2 undergoing the meditation practice for 8 weeks.

Baseline measurement details:

QUESTIONNAIRES: Each participant will be given a 1-item Visual Analogue Scale for stress (VAS), a 10 item Perceived Stress Scale (PSS), and a 9 item Pittsburgh Sleep Quality Index (PSQI) questionnaire. The VAS simply asks subjects to score how much stress they are feeling at that one moment in time on a 0-100 scale. The PSQI scores and assesses sleep quality and disturbances over a 1-month time interval and will be administered at the 4 week mark 1/2 way into the study as well as at pre and post intervention data collection events.

BLOOD PRESSURE: Blood pressure will be measured individually in a separate room to ensure confidentiality. The BP measurements will be administered using an Omron professional automatic blood pressure monitor (model number HEM 907X) to ensure comfort/safety and the accuracy of the reading. Also for accuracy of blood pressure measurements subjects will be asked to refrain from caffeine (coffee, tea or chocolate), cigarettes/nicotine, or exercise that morning until after measurements are taken and avoid alcohol the evening prior. One identified researcher will take all blood pressure reading and will be blinded to which subjects are part of the research or the control groups.

ELIGIBILITY:
Inclusion Criteria:

* Graduate student in the first year of the Doctorate of Physical Therapy (DPT) program at California State University, Northridge (CSUN)

Exclusion Criteria:

* Taking blood pressure or sleep medication; or already currently practicing a daily meditation.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure | 8 weeks
  Omron HEM 907XL professional automatic blood pressure monitor used at baseline and at 8 weeks post intervention
Change in Perceived Stress Survey Questionnaire | At baseline and at 8 weeks post intervention
  10-Item standardized survey tool for perceived stress level
Change in Sleep Hygiene utilizing PSQI survey | survey at baseline, 1 month and at conclusion of 8 weeks
  PSQI sleep survey administered 3 times during the study (baseline, 4 weeks and 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Beth J Phillips, PT, DPA, Principal Investigator — Full Professor
Locations (1):
- California State University, Northridge, Northridge, California, United States